CLINICAL TRIAL: NCT05646524
Title: A Phase II, Open-Label Study of NM8074 in Patients with Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Study of Efficacy and Safety of NM8074 in Adult PNH Patients Who Are Naive to Complement Inhibitor Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovelMed Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NM8074-PNH-105
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Intervention Model Description: 12 (18) patients will be divided into two cohorts of 6 (9) patients each. Patients will be dosed in parallel with either a 20 mg/kg NM8074 dose every two weeks for the entire duration of the treatment period or with an initial dose of 10 mg/kg NM8074 weekly for the first four weeks followed by the 20 mg/kg dose for the remainder of the treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): 6 subjects will receive an intravenous (IV) infusion of NM8074 at 20 mg/kg every two weeks.
  Interventions: Drug: NM8074
- Cohort 2 (Experimental): 6 subjects will receive an intravenous (IV) infusion of NM8074 at 10 mg/kg weekly for four weeks followed by a 20 mg/kg dose of NM8074 every two weeks for the remainder of the treatment period.
  Interventions: Drug: NM8074

INTERVENTIONS:
Drug: NM8074 — NM8074 will be administered as an intravenous infusion. Doses will be administered over a treatment period of 13 weeks.

SUMMARY:
This is a Phase II, open-label study designed to evaluate the safety, efficacy, and immunogenicity of NM8074 administered intravenously to adult patients with Paroxysmal Nocturnal Hemoglobinuria (PNH).

DETAILED DESCRIPTION:
The proposed study will enroll a planned number of 12 treatment naïve PNH patients with amaximum of 18 PNH patients who have been diagnosed with hemolytic anemia and meet the inclusion criteria. There will be 2 cohorts with 6 to 9 patients each. Patients in Cohort 1 will be administered NM8074 at 20 mg/kg intravenously (IV) every 2 weeks over the treatment period. Cohort 2 patients will be administered a dose of 10 mg/kg NM8074 weekly for 4 weeks followed by a 20 mg/kg dose of NM8074 administered via IV every 2 weeks for the remainder of the treatment period. This study will determine if NM8074 will provide the desired inhibition of the alternative pathway (AP).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years (males and females), weight ≥ 45 kg at the time of consent
* Confirmation of PNH diagnosis by flow cytometry evaluation of white blood cells (WBCs), with neutrophil, granulocyte and/or monocyte clone size of ≥10%
* Evidence of ongoing hemolysis
* ≥1 packed red blood cell (pRBC) transfusion within 12 months prior to screening
* Anemia (Hemoglobin ≤10.5 g/dL)
* Lactate dehydrogenase (LDH) level ≥ 1.5 times the upper limit of normal (xULN) during Screening
* All patients must be vaccinated prior to dosing with MenACWY Menactra® polysaccharide diphtheria toxoid conjugate vaccination against Neisseria meningitidis serogroups A, C, Y, and W-135 and MenB meningococcal serogroup B vaccine (Bexsero®). If the window of vaccination is short, then patients will be prophylactically treated with appropriate antibiotics
* Willing and able to understand and complete informed consent procedures, including signing and dating the informed consent form (ICF), and comply with the study visit schedule

Exclusion Criteria:

* History of bone marrow, hematopoietic stem cell, or solid organ transplantation
* History of splenectomy
* Participation in any other investigational drug trial within 5 elimination half-lives of enrollment, or within 30 days, whichever is longer
* Subjects currently or previously under other complement inhibitor treatments less than 3 months prior to study Day 1
* Participants with known or suspected hereditary or acquired complement deficiency
* History of currently active primary or secondary immunodeficiency
* Currently active systemic infection or suspicion of active bacterial, viral, or fungal infection within 2 weeks prior to first dose, or history of unexplained, recurrent bacterial infections
* Has a known history of meningococcal disease or N. meningitidis infection
* Patients on immunosuppressive agents or systemic corticosteroids less than 8 weeks prior to dosing
* Known medical or psychological condition(s) or risk factor that, in the opinion of the Investigator, might interfere with the patient's full participation in the study, pose any additional risk for the patient, or confound the assessment of the patient or outcome of the study
* Severe concurrent co-morbidities not amenable to active treatment, e.g., patients with severe kidney disease (chronic kidney disease (CKD) stage 4, dialysis)
* Subjects currently or previously under other complement inhibitor treatments less than 3 months prior to study Day 1
* Pregnant, planning to become pregnant, or nursing female subjects. Female partners of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must have a negative pregnancy test at screening and must agree to use highly effective methods of contraception during dosing and for 1 week after stopping the investigational drug
* Females who have a positive pregnancy test result at Screening or on Day 1
* Male patients and partners of child-bearing potential must agree to use contraceptives and male patients must agree to refrain from donating sperm for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Monitoring of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Study Day 105
  Adverse events will be graded according to the CTCAE v4.03. If the AE term is not described in the grading scales, the AE severity shall be reported according to the following:
  Grade I: Mild (awareness of sign or symptom, but easily tolerated)
  Grade II: Moderate (discomfort sufficient to cause interference with normal activities)
  Grade III: Severe (incapacitating, with inability to perform normal activities)
  Grade IV: Life threatening
  Grade V: Fatal
Number of Participants with Antidrug Antibodies (ADAs) to NM8074 | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in Hemoglobin (Hgb) Levels | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in Lactate Dehydrogenase (LDH) Levels | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in Number of Packed Red Blood Cell (pRBC) Transfusions | Up to Study Day 105
Percent Change from Baseline in Levels of Membrane Attack Complex (MAC) via Alternative Pathway (AP) of Complement Activity as Compared to Percent Change from Baseline in Levels of MAC via Classical Pathway (CP) of Complement Activity | Up to Study Day 105
Percent Change from Baseline in Levels of Complement Component C3b via Alternative Pathway (AP) of Complement Activity as Compared to Percent Change from Baseline in Levels of C3b via Classical Pathway (CP) of Complement Activity | Up to Study Day 105

SECONDARY OUTCOMES:
Change from Baseline or Percent Change from Baseline in Reticulocyte Count | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in Bilirubin Levels | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) Survey Assessed via the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale, Version 4. | Up to Study Day 105
  The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue with a 7-day recall period. Items are scored on a 0 - 4 response scale ranging from "Not at all" to "Very much so". All items are summed to create a single fatigue score with a range from 0 to 52 with a better quality of life indicated by a higher score.
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) Survey Assessed via the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 Scale (QLQ- C30), Version 3.0. | Up to Study Day 105
  All EORTC QLQ-C30 scales and single-item measures range from 0 to 100. This includes 3 symptom scales (fatigue, pain, nausea and vomiting), 5 functional scales (physical, role, cognitive, emotional, and social), single-item questions addressing symptoms like insomnia, dyspnea, loss of appetite, and others that are commonly reported by cancer patients, and the perceived financial impact of the disease. A higher score is associated with a greater quality of life for global health status.
Changes in plasma concentration of NM8074 | Up to Study Day 105
Maximum plasma concentration (Cmax) | Up to Study Day 105
Time corresponding to Cmax (tmax) | Up to Study Day 105
Area Under the Drug Concentration-Time Curves (AUC0-t) | Up to Study Day 105

OTHER OUTCOMES:
Change from Baseline or Percent Change from Baseline in Complement Component Factor B Levels | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in Haptoglobin Levels | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in Platelet Count | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in PNH Cell Clone Size | Up to Study Day 105
  Clone size will be measured via fluorescein-labeled proaerolysin (FLAER) staining of WBCs (granulocytes and monocytes)
Change from Baseline or Percent Change from Baseline in C3b Deposition on PNH Cells | Up to Study Day 105
  Loading of C3b on erythrocytes will be evaluated using flow cytometry
Change from Baseline or Percent Change from Baseline in Levels of Membrane Attack Complex (MAC) via Classical Pathway (CP) of Complement Activity | Up to Study Day 105
Change from Baseline or Percent Change from Baseline in Levels of Complement Component C3b via Classical Pathway (CP) of Complement Activity | Up to Study Day 105

IPD SHARING:
Plan to Share IPD: No